CLINICAL TRIAL: NCT00166218
Title: Evaluation of Near-infrared Spectroscopy for Non-invasive Monitoring of the Ambulatory Single Ventricle Patient
Brief Title: NIRS Monitoring in the Ambulatory Single Ventricle Patient
Status: Terminated | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, William T. Mahle, MD, Principal Investigator, Emory University
Other Study IDs: 0793-2003
Record Dates: First submitted 2005-09-13; First posted 2005-09-14 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Ambulatory Children With Single Ventricle
Keywords: pediatrics; cardiac defects
MeSH Terms: interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Device: near-infrared spectroscopy

SUMMARY:
The normal heart has four chambers. There are two upper (or filling) chambers and are called the atrium. There are two lower (or pumping) chambers and are called the ventricles. One of the ventricles pumps blood to the lungs to get oxygen. This oxygenated blood is returned to the heart then pumped to the rest of the body by the other ventricle.

Sometimes babies are born with heart defects that only allow one of the lower chambers (ventricle) to work properly. This means that the one ventricle must pump blood to both the lungs and to the rest of the body. Babies born with this defect must undergo multiple surgeries, the first of which is usually done during their first week of life.

There is a machine that is FDA approved that can measure how much oxygen is delivered to the brain. This non-invasive (outside the body) machine uses Near-infrared spectroscopy (NIRS), which is similar technology used in pulse oximetry and is routinely used to measure the level of oxygen in blood. At Children's Healthcare of Atlanta, we typically place the NIRS machine on the baby in the Cardiac Intensive Care Unit immediately after their first surgery to monitor oxygen delivery to the brain. The monitor has proven to be accurate in this situation.

We now want to know if we can use this monitor to assess oxygen delivery to the brain before and during a routine heart catheterization prior to the child's second surgery. Once consent is obtained, we will place a probe on the child's forehead during the pre-catheterization visit and obtain readings for 5 minutes. The probes are about the size of a quarter and are self-stick (they look like the kind of leads used to measure the babies heart rate [EKG]). The machine will be disconnected for the rest of the Pre-catheterization visit, however the probes will stay on the child's forehead. Once the child is in the catheterization suite, the machine will be reconnected. A sheath or hollow tube is routinely placed in a blood vessel in the child's neck or groin for the catheterization. The doctor would place a special catheter in this sheath that measures oxygen levels in blood continuously. This monitor would be calibrated by using the results of a blood sample that is routinely drawn from the child's IV. During the same sampling, an additional 2cc's of blood would be collected to measure the lactate level. The lactate level is an indicator of how well the child is using oxygen. Once this monitor is calibrated, data will be collected for 5 minutes to compare it with the NIRS machine. The special catheter will be removed after the 5-minute time period, and the catheterization will proceed as usual. The NIRS probes will stay on the child's forehead during the entire catheterization with the data documented. At the end of the catheterization, the probes will be removed.

DETAILED DESCRIPTION:
The study will be a prospective evaluation of all single ventricle patients as they undergo their routine cardiac catheterization prior to second stage palliation. Upon arrival to the pre-catheterization area, NIRS probes will be placed on the child's forehead and data along with vital signs will be collected at initial placement, 3 minutes and at 5 minutes. The monitor will be disconnected as the routine pre-catheterization procedures proceed.

Once the child is in the catheterization suite, the monitor will be reconnected and the routine catheterization procedures will proceed. After the standard sheath for catheterization is placed in the child, a routine superior vena cava saturation (COOX) will be drawn and the NIRS reading along with routine vital signs will be documented. At the same time the routine saturation is drawn, an additional 2ccs of blood will be drawn for a lactate level. At 3 and 5 minutes after the routine saturation, a COOX will be drawn and the NIRS reading along with vital signs will be documented. The catheterization will continue as usual. At the end of the case, a final NIRS reading and vital signs will be documented prior to the removal of the probes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with single ventricle anatomy undergoing routine, elective cardiac catheterization prior to second stage palliation.
2. Parental consent to participate in the study -

Exclusion Criteria:

1. Admission to the Intensive Care Unit or intubation prior to catheterization
2. Emergent catheterization -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2004-02; Study Completion 2005-02

CONTACTS AND LOCATIONS:
Overall Officials: Robert Vincent, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia, United States

REFERENCES:
- [Background] Kurth CD, Steven JL, Montenegro LM, Watzman HM, Gaynor JW, Spray TL, Nicolson SC. Cerebral oxygen saturation before congenital heart surgery. Ann Thorac Surg. 2001 Jul;72(1):187-92. doi: 10.1016/s0003-4975(01)02632-7. PMID 11465176